CLINICAL TRIAL: NCT03562351
Title: Seizure Rescue Medication: Caregiver Education in a Simulation Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Tobias Loddenkemper, Associate Professor, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P00027241
Record Dates: First submitted 2018-03-06; First posted 2018-06-19 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Status Epilepticus
MeSH Terms: conditions — Status Epilepticus

STUDY DESIGN:
Intervention Model Description: The investigators will implement an intervention jointly with our simulation program to determine the most effective training model: verbal instructions, instructional video, or use of a mannequin. Caregivers will undergo a training curriculum, and 90 caregivers (30 assigned to each educational model) will be matched into three groups and assigned to participate in one of three educational models in the SIM Center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Verbal Instructions on use of RM (Experimental): Caregivers will undergo an educational intervention with typical training with verbal instructions and use of a rectal diazepam trainer.
  Interventions: Other: Verbal Instructions Educational Intervention
- Video on use of RM (Experimental): Caregivers will undergo an educational intervention with training by watching an instructional video regarding rescue medication administration
  Interventions: Other: Video Educational Intervention
- Mannequin on use of RM (Experimental): Caregivers will undergo an educational intervention with training by use of a mannequin to practice administering the rescue medication
  Interventions: Other: Mannequin Educational Intervention

INTERVENTIONS:
Other: Verbal Instructions Educational Intervention — Caregivers will undergo training with verbal instructions
  Arms: Verbal Instructions on use of RM
Other: Video Educational Intervention — Caregivers will undergo training with an educational video
  Arms: Video on use of RM
Other: Mannequin Educational Intervention — Caregivers will undergo training with a mannequin
  Arms: Mannequin on use of RM

SUMMARY:
1. Design an educational quality improvement program to assess the most effective educational approach on caregiver seizure RM application. The investigators hypothesize that this educational program will improve caregiver comfort, knowledge of emergent seizure care, and time to medication application.

Specifically, the aims include:

1. Create an educational video reviewing RM administration
2. Develop and validate a simulation training model/mannequin for rectal diazepam administration
3. Expand training to other seizure RMs (e.g. intranasal midazolam, buccal lorazepam) and transition the most effective educational model back to the clinics/bedside to standardize caregiver teaching throughout the department/hospital

DETAILED DESCRIPTION:
The investigators will implement an intervention jointly with a simulation program to determine the most effective training model: verbal instructions, instructional video, or use of a mannequin. Caregivers will undergo a training curriculum, and 60 caregivers (20 assigned to each educational model) will be matched into three groups and assigned to participate in one of three educational models in the SIM Center. Pre-and post-training questionnaires will be distributed to assess provider knowledge and comfort level. Scoring of caregiver technique administering rectal diazepam to a mannequin and time to RM administration will be obtained to compare between the three educational arms of the study. Thirty additional patients (10 per group) will not receive an assessment of caregiver technique administering RM to the mannequin prior to the educational intervention to control for exposure to the mannequin. Ultimately, the most effective educational method in this simulation pilot study will be expanded to other RM types (e.g. intranasal midazolam, buccal lorazepam), standardized, and brought back to the clinics/bedside throughout the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Adult caregivers of patients with epilepsy followed at BCH with the following:

   1. At least one seizure >5 minutes
   2. Prescription for rectal diazepam rescue medication
   3. Admission for seizure/neurologic problem or neurology/epilepsy clinic visit during the enrollment period
2. Adult caregivers of patients without epilepsy

Exclusion Criteria:

1. Adult caregivers of epilepsy patients without a rectal diazepam prescription
2. Non-English-speaking caregivers

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Change in Time to RM Administration | Baseline and 30 minutes post-intervention
  As determined by time to administer RM to mannequin

SECONDARY OUTCOMES:
Change in "RM Score" | Baseline and 30 minutes post-intervention
  "RM Score" ("Rescue Medication Score") assessing caregivers' ability to administer RM with proper technique before/after training. This score will determine if caregivers were able to independently give the medication or if they required a prompt at any step. There is no maximum score, but 1 point will be given for every required prompt such that 0 is a perfect score and higher scores reflect requiring more prompts to administer the medication.
Change in Caregiver Level of Knowledge of Medication Name | Baseline and 30 minutes post-intervention
  Caregiver will be asked to provide medication name on a questionnaire.
Change in Caregiver Level of Knowledge of When to Give Medication | Baseline and 30 minutes post-intervention
  Caregiver will be asked to provide time at which medication is to be given on a questionnaire.
Change in Caregiver Level of Knowledge of Route of Medication Administration | Baseline and 30 minutes post-intervention
  Caregiver will be asked to provide route of medication administration on a questionnaire.
Change in Caregiver Level of Knowledge of Medication Side Effects | Baseline and 30 minutes post-intervention
  Caregiver will be asked to provide medication side effects on a questionnaire.
Change in Caregiver Level of Comfort | Baseline and 30 minutes post-intervention
  Caregiver level of comfort with administration as determined by the pre- and post-questionnaires. Caregivers will report level of comfort before and after training based on a 4-point scale (very uncomfortable, somewhat uncomfortable, somewhat comfortable, very comfortable)
Change in Caregiver Feeling of Ease with Administration | Baseline and 30 minutes post-intervention
  Caregiver level of ease with administration as determined by the pre- and post-questionnaires. Caregivers will fill out the short-form State-Trait Anxiety Inventory (STAI-6) on a 4-point scale (not at all, somewhat, moderately, very much)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No